CLINICAL TRIAL: NCT07309523
Title: The Force Frequency Relationship in Heart Failure: an Expression of a Metabolic Problem Driving Adverse Remodelling?
Brief Title: The Force Frequency Relationship in Heart Failure and Diabetes Mellitus: a Metabolic Aetiology?
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Klaus K Witte, MD, Senior Lecturer in Cardiology, University of Leeds
Other Study IDs: 2024-NCT17
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Diabetes (DM)
Keywords: Force frequency relationship, heart failure, diabetes mellitus, Treppe
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skeletal muscle, blood, fat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HFrEF without DM: People with heart failure due to reduced ejection fraction
- HFrEF with DM: People with heart failure due to reduced ejection fraction who also have diabetes mellitus
- No HF, no DM: People without heart failure who also do not have diabetes mellitus
- No HF but with DM: People without heart failure but who do have diabetes mellitus

SUMMARY:
The present investigation is a non-randomised, observational study involving an unselected but highly phenotyped cohort of patients undergoing pacemaker or defibrillator implantation from whom a small sample of fat and muscle will be taken from the operation site, and, in a subgroup, from the thigh muscle. A sample of blood wil also be taken from the vein of the heart, a peripheral vein and the artery at the wrist during the procedure at different heart rates and pacing modes, to describe how heart rate and heart contraction power relate to cardiac and peripheral metabolism.

The coded blood and tissue samples and anonymised clinical data will be stored in a Human Tissue Authority-approved freezer until analysis.

Following the procedure, during routine visits, patients' left ventricular force frequency relationship will be assessed using cardiac ultrasound and a non-invasive cardiac monitor to further phenotype the severity and progression of their heart function over 6 months. For most patients, their involvement will end at that point although they will be monitored through electronic health records on an annual basis from that point forward for up to 5 years after the end of the study (for up to ten years after that point) to gain information on the prognostic value of the metabolic and haemodynamic testing.

The present investigation will allow the investigators to advance the understanding of heart-muscle crosstalk with the goal of developing targeted interventions that could open new treatment avenues.

DETAILED DESCRIPTION:
RESEARCH QUESTION Hypothesis: The abnormal cardiac force-frequency relationship (FFR) and peripheral autonomic activation are the result of cardiac and peripheral metabolic abnormalities.

Fundamental aims: to determine whether impaired metabolism is a mechanism underlying the failing FFR in patients with heart failure and to determine whether diabetes mellitus is a contributing factor to the development of heart failure through its adverse effect on metabolism reflected in an abnormal FFR.

Secondary aims - this project will provide answers to a series of important questions through a single protocol which are potentially of direct and longer term importance to patients:

1. What metabolic pathways are abnormal in people with heart failure, diabetes mellitus and both?
2. What is the relationship between skeletal muscle metabolic abnormalities and those of the myocardium?
3. Can we identify using metabolomics, a substrate or compound that underlies the metabolic abnormalities?
4. What is the effect of diabetes mellitus on cardiac (glucose) and peripheral metabolism at rest and with increased heart rate?
5. Is cardiac metabolism abnormal at higher heart rates despite adequate perfusion?
6. Is abnormal cardiac metabolism related to that of the peripheral muscles?
7. Does this 'cross-talk' have a negative influence on the FFR and how does this relationship change with increased heart rate?
8. Can the improved FFR with CRT be explained by improved cardiac metabolism across the entire heart rate range?
9. Is peripheral autonomic activation at higher heart rates reflected in higher activation of cardiac sympathetic tone in HFrEF?
10. Do the laboratory data about muscle, fat and metabolomics relate to clinical variables, response to therapy and prognosis?
11. Do the haemodynamic responses to heart rate increase predict outcomes following pacemaker insertion?

STUDY DESIGN AND SETTING This will be a UK-based, unblinded, observational, mechanistic study carried out in patients receiving a pacemaker device as standard of care.

PARTICIPANT RECRUITMENT AND ELIGIBILITY CRITERIA Identification, approach and consent: Patients with and without heart failure as well as with and without type 2 diabetes mellitus receiving a clinically indicated pacemaker implantation will be approached. The selection of patients for device therapy is based on the current European guidelines on heart failure and also the European Guidelines on Pacemaker Therapy from the European Society of Cardiology (ESC) 2021. The diagnosis of T2DM is made based on HbA1c, fasting glucose, existing antidiabetic medication and/or a pathological glucose tolerance test. Patients with impaired glucose tolerance, as a precursor to overt T2DM, will also be included. In study participants of childbearing age, pregnancy is routinely excluded for clinical reasons before device implantation due to the potential risk of exposure to X-rays.

The clinical teams will approach, and the research team will follow-up these approaches, aiming for an estimated 180 patients, to achieve 160 participants (40 with CHF and DM, 40 with CHF but without DM, 40 without CHF but with DM, and 40 with neither CHF nor DM).

Participants will not be paid for participation, although reasonable travel costs will be refunded according to guidelines laid out by INVOLVE.

STUDY CLINICAL PROCEDURES:

Baseline visit (pre-implantation): Patients will be approached by the study team only after their clinical team has identified that they are suitable and interested. Patients will be offered an information sheet and be given a week to read and consider it. They will then receive a telephone call from the study nurse or doctor prior to attending the baseline visit to check if they are interested and to answer any outstanding questions.

If they agree to participate, they will attend for their baseline visit around one week prior to the day of the procedure. This visit will be combined with the pre-assessment visit for the pacemaker device implant to save them a second hospital attendance.

At the baseline visit the following tests will be done:

1. Demographics, co-morbidities, medical therapies, height, weight: These will also be entered on the pre-assessment form for the pacemaker procedure.
2. Two quality of life questionnaires (the Kansas City Cardiomyopathy Questionnaire and EQ5D-5L) (research activity)

2) Frailty assessment: Frailty is an important risk factor for adverse outcomes in heart failure. One component contributing to frailty is muscle strength. Hence, we will include an assessment of frailty known as the clinical frailty scale (CFS). This is not a questionnaire and requires no input from the patients and is routinely collected for the pacemaker procedure. They will also complete a questionnaire specific for sarcopenia to improve the identification muscle loss (research activity).

3) Echocardiography: This is routinely in use in research projects in Leeds. In this protocol it would be a research activity unless not done clinically in the last 6 months, in which case it would have been repeated prior to the pacemaker implantation. All participants will undergo complete echocardiography with two-dimensional grayscale and tissue Doppler images recorded in two- and four-chamber. The images are stored in the "Echopac" digital imaging system and analyzed offline (GE, Milwaukee, WI, USA). This analysis includes a calculation of LV end-diastolic and end-systolic volumes using the biplane disk method (modified Simpson method). The frame at the R wave is taken as end diastole and the frame with the smallest LV volume is taken as end systole. The LV end-systolic volume (ESV) index (ESVi) is calculated as ESV/body surface area (BSA) in each phase. Each measurement is averaged from three beats. BSA is calculated using the Mosteller equation. Our data to date have confirmed good reproducibility. This method of LV volume calculation is not only widely used and accepted, , but the key variable is the ESV, which has a particularly high reproducibility.

4) An exercise ECG with metabolic gas analysis (cardiopulmonary exercise test) will be performed depending upon pacemaker indication. This is a common functional test established in the clinic to assess a patient's performance. The patient will walk continuously on a treadmill until exhaustion. The aim is to evaluate the patient's maximum performance. As part of the examination, blood pressure, pulse and oxygen saturation will be measured at three minute intervals. A stress ECG is usually carried out to assess progress before and after therapy (in this case CRT implantation) and is normally therefore carried out on an outpatient basis before CRT implantation and 6 months afterwards. For those receiving a pacemaker for intermittent bradycardia this will be done approximately 6 weeks after implantation of the pacemaker system to avoid the confounding of a bradycardia.

5) Handgrip strength (research activity): Lower handgrip strength is a marker of adverse outcome in CHF,[ ] and we have previously demonstrated a relationship to exercise capacity. As a non-invasive marker of skeletal muscle function each will be asked to perform maximal handgrip strength assessment using a standard handgrip dynamometer (Jamar). This will be recorded as the best of three attempts on the non-dominant arm.

6) Bioimpedance to assess lean mass (research activity): Higher lean muscle mass and higher fat mass are associated with better outcomes in people with heart failure. Body composition assessment may help define and clarify the obesity paradox in heart failure where, despite a higher rate of heart failure in obese people, worse rates of diabetes (an adverse factor in CHF) and lesser exercise tolerance, obesity is associated with better outcomes in cohort studies of people with prevalent heart failure. A portable bioelectrical impedance device will be used to assess the proportion of muscle and fat.

7) Blood tests for kidney function, glucose levels and HbA1c (routine clinical activity but blood also taken for research purposes and results used for research database): Those data collected for this study that are relevant to clinical care (peak oxygen consumption and echocardiography) including this exercise test will be added to the medical record to save the patient multiple exercise tests.

During the procedure: The device implantation will be performed according to standard protocols, within two weeks of the preassessment.

Once the routine implantation of the leads has taken place, the participant will be asked to confirm that they remain comfortable and happy to continue with the study procedures of heart rate adjustment and blood sampling.

Patients receiving a pacemaker routinely receive a venous cannula to allow provision of drugs including antibiotics and fluids.

1. Optional thigh muscle biopsy (research procedure): Prior to the start of the pacemaker procedure, a thigh muscle biopsy will be done in a subgroup of patients. This will be included as an optional procedure in those participants that have agreed and provided consent to this additional procedure. Many previous studies that have assessed skeletal muscle function in both CHF patients as well as numerous other populations have used muscle biopsies from the vastus lateralis muscle of the thigh. This particular muscle is considerably more susceptible to the effects of training and detraining. Therefore in order to establish the differences in patients that are attributable to detraining as opposed to systemic differences, a biopsy will be taken from both muscles (pectoralis major and vastus lateralis).
2. Invasive arterial monitoring (research procedure): In patients with HF, an arterial pressure catheter is often placed for invasive blood pressure monitoring (usually radial artery). In addition, there is one peripheral venous access as standard. In patients undergoing a standard pacemaker implantation, this would be a study-related procedure.
3. Invasive haemodynamics (research procedure): In addition, in a subgroup of people in each group (n=40 in total), using the venous access required for the pacemaker implantation, we will pass a catheter through the heart into the pulmonary artery to measure the pressures 'behind' the left ventricle (the main pumping chamber). This is a routine procedure in the assessment of severe heart failure. The measurement of pulmonary artery and left atrial pressure in this way would represent a research procedure for those people having a pacemaker that do not have heart failure.
4. Non-invasive cardiac monitoring (research procedure): Cardiac output and pulse pressure will be assessed through small blood pressure cuffs on patients' fingers throughout the procedure and specifically at different heart rates.
5. Pectoralis muscle and subcutaneous adipose tissue sampling (research procedure): During creation of the pacemaker pocket, muscle and fatty tissue are exposed and three samples of muscle and three samples of fatty tissue each less than 2mm x 2mm will be taken and immediately frozen in liquid nitrogen. The sampling is painless.
6. Lead implantation (routine clinical activity): The cardiac leads are inserted into the heart via the subclavian vein. A lead is first implanted in the right ventricle and, if indicated, a lead is placed in the right atrium.
7. Coronary sinus cannulation (research/standard activity): To insert the CS lead for CRT pacemaker implantation, the coronary sinus is routinely first cannulated using a guide catheter, through which blood can be taken easily. The coronary sinus represents the venous drainage system of the heart and a comparison of the coronary sinus blood ("output") with the arterial blood ("input") allows conclusions to be drawn about cardiac metabolism. This method for studying cardiac metabolism is recognized and has been used by numerous other groups. Most recently this technique has been used to describe the persistent metabolic flexibility of the heart despite CHF.

   For patients without an indication for CRT, coronary sinus cannulation would be study-based and follow exactly the same protocol as for patients with HF. In less than 0.5% of coronary sinus intubations (1 in 200), a dissection of the vein can occur (similar to a bruise on the hand when a venous cannula is inserted). In patients indicated for a normal pacemaker, this type of dissection would have no clinical consequences because it heals immediately within a short period of time and does not stop the implantation of the currently indicated pacemaker.

   X-ray dose size: The average published acceptable effective dose for a routine normal pacemaker implantation is 1.1-1.7mSv. , The CI (KKW) routinely collects these data for their own governance processes. In >1500 consecutive normal pacemaker implantations the fluoroscopy time for a normal pacemaker implantation (performed by the CI) is on average 4 minutes, corresponding to an average dose area product of 435cg/cm2 and an average effective dose of 0.57mSv.

   There are no published recommended dose ranges for cannulation of the coronary sinus since the relevant values are for the entire coronary sinus lead placement procedure (which includes cannulation). The CI has prospectively collected the time taken to achieve CS cannulation in the last 11 clinically indicated cases of CRT implantation. CS cannulation was achieved in 58 (range 21-103) seconds with an average effective dose of 0.18 (0.06-0.35) mSv. Hence, the effective dose for patients receiving a standard pacemaker who participate in this study, despite the addition of a study-related coronary sinus cannulation, is likely to be below the published effective dose for a standard pacemaker implantation. Hence, the probability of any radiation-induced tissue damage or complication is therefore very low.

   X-ray contrast dose: Usually, around 10-15ml of contrast is required to achieve coronary sinus cannulation. This amount of contrast is very unlikely to cause kidney damage. A known allergy to contrast media and an eGFR<20 are exclusion criteria.
8. Blood collection at rest (research activity): After cannulation of the coronary sinus, coronary sinus blood will be collected for the study via the guide catheter and at the same time arterially via the pressure catheter and peripheral-venous via an indwelling venous catheter. The blood collection will require no more than 1-2 minutes.
9. Blood collection at higher HR (to assess the FFR)(research activity): Using the implanted leads, the heart rate is then increased in three phases to 75, 100 and 125 beats per minute. This ensures that most participants have a heart rate two levels below that critical heart rate and one above it. Blood is taken again at each heart rate.

Total volume of blood: A total of around 50 ml more blood will be taken than would normally be the case during a pacemaker implantation.

Completion of the procedure (routine procedure): The operation will then be carried out as follows planned and the immediate postoperative care will be carried out according to the usual care with normal pain relief and blood pressure checks.

Predischarge assessment (routine assessment): A formal pacemaker check and echocardiogram will be undertaken pre discharge. This assessment will include a non-invasive assessment of the cardiac output using the Finapress device and an assessment of the FFR as previously described which would both be research procedures. The leg wound will be checked if a thigh muscle biopsy has been done.

Medium-term follow-up: After 4-6 weeks participants will return for their routine check-up appointment. This will include an echocardiogram and FFR assessment (both of which would be research activity) and will replace their usual pacemaker appointment. Those who did not have an exercise ECG preoperatively will have one performed (research activity) and all patients will complete the two questionnaires (research activity). Bioimpedance and handgrip strength measurements (research activity) will also be undertaken at this point.

Long-term follow-up: As part of routine pacemaker check at 6-7 months after the implantation, an echocardiographic follow-up (routine clinical activity) and interrogation of the pacemaker will include a review of the medications and an assessment of frailty as previously (research activity). Bioimpedance and handgrip strength measurements (research activity) will also be undertaken at this point.

Prognostic relevance of the FFR (research activity): Electronic health records will determine vital status, collect data on hospitalization, cardiovascular events (heart attack, stroke, cardiac decompensation, cardiac arrhythmias, assistive devices, heart transplant) and death up to 5 years after the end of the recruitment phase such that some participants might be followed for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Guideline-compliant, clinical indication for pacemaker implantation
* Age >18 years
* Ability to provide written informed consent
* Persons who are legally competent and mentally able to follow the instructions of the study staff

Exclusion Criteria:

* Anemia Hb <8 mg/dl
* Patients with acute infectious diseases (e.g. pneumonia)
* Patients with heart failure due to sepsis
* People with acute myocardial ischemia, which is manifested, for example, by angina pectoris or ECG changes under stress
* Patients with acute liver or kidney failure
* Pregnant and breastfeeding women
* People who are institutionalized on official or court orders
* People who are dependent or employed by the sponsor or investigator
* Taking study medication (of an investigational drug) 30 days before the start of the study
* Known contrast allergy or eGFR <20ml/min/1.73m2
* Pregnancy not excluded by bedside pregnancy test in premenopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People having an implantable cardiac device procedure
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-08-30 (Estimated); Study Completion 2034-08-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between FFR and cardiac metabolomics | At baseline
  Is cardiac metabolism in patients with diabetes and diabetes with heart failure as assessed by mass spectrometry-based metabolomics and lipidomics abnormal at higher heart rates and is the degree of the impairment correlated with the heart rate at which peak contractility occurs?

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised dataset
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after the publication of the main results
Access Criteria: By an email to the PI access to the file through a secure site.